CLINICAL TRIAL: NCT07156214
Title: Pathogenic Insights and Search for Biomarkers in RFC1-ataxia/CANVAS: a Model to a Deeper Understanding of Molecular Mechanisms Underlying Late-onset Neurodegeneration
Brief Title: Pathogenic Insights and Search for Biomarkers in RFC1-ataxia/CANVAS
Acronym: INSIDE-CANVAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6336
Record Dates: First submitted 2025-07-29; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-07

CONDITIONS: CANVAS Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CANVAS patients (Other): Patients with molecular diagnosis of RFC1-ataxia
  Interventions: Other: Assessment of markers of oxidative stress in peripheral blood samples
- Healthy controls (Active Comparator): Partners of patients with RFC1-ataxia
  Interventions: Other: Assessment of markers of oxidative stress in peripheral blood samples

INTERVENTIONS:
Other: Assessment of markers of oxidative stress in peripheral blood samples — Participants will perform serial blood samples at interval of 12 months to compare levels of markers of oxidative stress
  Other Names: Characterization of mitochondrial function on fibroblasts derived from skin biopsies available at our Laboratory for research purposes and generation of iPS cells

SUMMARY:
CANVAS (Cerebellar Ataxia, Neuropathy, Vestibular Areflexia Syndrome), also referred to as RFC1-ataxia, is a recently molecularly characterized neurodegenerative disorder caused by a biallelic expansion of an AAGGG pentanucleotide repeat in intron 2 of the Replication Factor C subunit 1 (RFC1) gene.

This adult-onset condition presents with a variable combination of cerebellar ataxia, peripheral neuropathy, and vestibular dysfunction. Currently, limited data are available regarding its natural history and the molecular mechanisms by which this dynamic mutation leads to neurodegeneration of selective neuronal populations.

Given that recent literature identifies RFC1/CANVAS as a relatively common genetic cause of late-onset ataxia, elucidation of its underlying pathogenic mechanisms may offer insights into the molecular pathways implicated in more prevalent late-onset neurodegenerative diseases, such as Parkinson's disease and Alzheimer's disease.

DETAILED DESCRIPTION:
The research proposal recognizes as the primary aim to evaluate and compare the sensitivity of individual validated clinical rating scales in assessing global disease severity and/or progression in a cohort of RFC1-ataxia patients Secondary aims are i) to identify novel potential circulating biomarkers in RFC1-ataxia by testing a cohort of RFC1-ataxia patients vs controls and ii) to establish and study patient-derived cell models to get insight about pathogenesis of RFC1-ataxia, particularly concerning mitochondrial function.

For these purposes, a longitudinal assessment of a study cohort of genetically determined RFC1- ataxia patients ( intention to treat 25 pts) will be carried out.

Based on the involvement of cerebellar and proprioceptive systems in RFC1-ataxia, the following clinical rating scales have been selected: Scale for the Assessment and Rating of Ataxia (SARA) , International Cooperative Ataxia Rating Scale (ICARS), SEnsory Ataxia Rating Scale (SEARS) , Berg Balance Scale (BBS) , and Tinetti Assessment Tool . Vestibular symptoms will be assessed by Dizziness Handicap Inventory questionnaire (DHI).

For statistical analysis regarding clinical severity, at T0 (baseline) RFC1- patients will also undergo:

1) neurophysiological studies: EMG and nerve studies, motor and sensory evoked potentials recorded at the four limbs; 2) vestibular function assessment by video head-impulse-test. Collected data will also include: age at onset (AAO) of symptoms, age at enrollment (AAE), disease duration (DD); presence of unexplained cough and/or swallowing disturbances; 3T brain and spinal cord MRI. Statistical analysis will be performed by Pearson's correlation tests . Global and item scores for each scale will be also correlated with DD, disability stage estimated by the SPATAX disability score (0: no functional handicap, 1: no functional handicap but signs at examination, 2: mild, able to run, unlimited walking, 3: moderate, unable to run, limited walking without aid, 4: severe, walking with one stick, 5: walking with two sticks, 6: unable to walk, requiring a wheelchair, 7: confined to a bed), and other major diagnostic findings individually contributing to motor disability ( i.e. neuropathy, vestibulopathy, cerebellar atrophy) .

For the second aim, blood samples will be collected from the RFC1- ataxia cohort and a cohort of age-and sex matched healthy controls enrolled to this purpose for the assessment of a panel of circulating biomarkers of oxidative stress (OS) and neurofilament light chain (Nfl), at both T0 (baseline visit) and T1 (one-year follow-up visit). Blood samples will be processed to obtain serum, plasma and RNA. For serum analyses, 9 cc of blood in Vacuette (CAT serum sep clot activator) tube will be drawn, centrifuged within 1 hour, aliquoted in multiple 50 uL aliquots, and stored at -80°C. For plasma analyses, 9 cc of blood will be drawn into EDTA tubes and, after 30' at room temperature, will be centrifuged and aliquoted in 50 uL aliquots and stored at -80°C. Lastly, venous blood will be drawn into one 10 ml BD Vacutainer tube with EDTA, and total RNA will be extracted from leukocytes and reverse-transcribed into cDNA, that will be stored at -80°C. All the samples collected will be stored, then, at the end of the collection period, will be shipped and examined simultaneously in duplicate to avoid freeze-thaw cycles, using an external service (laboratory of Molecular Medicine of the Bambino Gesù Hospital, Rome) The oxidative stress panel will include: expression of the transcription factor NRF2 (Nuclear factor erythroid 2-related factor 2) analyzed by Real Time-PCR. NRF2 regulates many cytoprotective pathways through the activation of antioxidant defenses, inhibition of inflammation, improvement of mitochondrial function, and maintenance of protein homeostasis. Of note, changes in this pathway have been associated to neurodegenerative diseases associated with mitochondrial dysfunction, in particular Friedreich ataxia. Serum markers related to antioxidant response include: glutathione peroxidase, reduced glutathione (GSH) and oxidized glutathione (GSSG), and glutathione metabolism (gamma-glutamylcysteine ligase, glutathione reductase) measured in sera by spectrophoto-fluorimetric assays and enzyme-linked immunosorbent assay (ELISA).

NfL levels will be assessed by Ella automated immunoassay. Results obtained in both RFC1 patients and controls will be statistically compared by Mann Whitney U-test (BM SPSS Statistics for Windows, Version 24.0. Armonk, NY) to test if any biomarkers would be significantly different in RFC1 patients, thus potentially representing a disease biomarker. In case of positive results, to assess the role as a disease severity marker, their levels will be correlated both with global and item scores of the clinical rating scale being the most sensitive among those tested in the cohort. Also, their levels at T0 and T1 will be compared in CANVAS -RFC1 patients vs controls, for evaluating their potential role as disease progression biomarker.

Another secondary aim consists in the deep characterization of mitochondrial function in RFC1 patient-derived fibroblasts, and the establishment of Induced Pluripotent Stem (IPSc) cell lines for future research Previous studies conducted on CANVAS patients' tissues apparently showed normal protein and transcripts levels of RFC1, however studies concerning a putative RFC1 function in mtDNA mantainence (replication and/ or repair) and related OXPHOS defect have not been performed so far. To this purpose, patients- and controls-derived primary fibroblasts (PF) (8 distinct RFC1 patients and 8 matched healthy controls) will be analyzed in parallel. RFC1 protein and mRNA levels will be quantified through Western blot (WB) and quantitative (q)PCR, respectively on total protein and RNA extracted from cell lysate to assess the presence of any significant reduction in RFC1 protein or transcript levels between CANVAS pts and controls.

Studies on oxidative stress and mitochondrial function: preliminary data of the investigators support that mitochondrial dysfunction might play a role in the pathogenesis of RFC1-ataxia, as the electron microscopy revealed the presence of clear mitochondrial abnormalities in RFC1 patients' derived fibroblasts ( two distinct cell lines).

To verify this hypothesis ,mitochondrial function will be assessed in RFC1 and controls fibroblasts by different approaches:

i) the presence of mitochondrial dysfunction is often associated with alterations either in dynamics, morphology and ultrastructure of mitochondria. These features will be investigated by confocal and transmission electron microscopy (TEM). For in vivo cell imaging, cells will be stained with Mitotracker Red, and Hoechst (nuclear probe). Images will be then captured by using a A1 confocal microscope, and image analysis will be performed using a specific software (Nikon Instruments). Cells will be scored into three categories: filamentous, intermediate, and fragmented mitochondria. Mitochondria ultrastructure will be analyzed on ultrathin fixed cells sections by a Tecnai G2 (FEI) TEM .

ii) mitochondrial dysfunction can also activate mitophagy, with consequent decrease of the mitochondrial mass contributing to cell energy defect. Mitochondrial mass will be assessed by immunoblot of porin and TOM20, two mitochondrial proteins index of mitochondrial mass. As additional indexes, both citrate synthase activity, a mitochondrial matrix enzyme, by spectrophotometry, and total mtDNA copy number by qPCR will be measured .

iii) to highlight presence of impaired OXPHOS process in RFC1 cells, fibroblasts will be forced to utilize mitochondrial OXPHOS to synthesize ATP by substituting galactose to glucose in culturing medium. The entry of galactose into glycolysis occurs at a significantly lower rate than glucose. So, RFC1 and control fibroblasts will be cultured in DMEM containing either glucose or galactose as main energy substrate for up to 72 h, and cell growth will be analyzed. To deeply investigate OXPHOS, oxygen consumption rate will be measured in digitonin-permeabilized cells (OCR) under state 4, state 3 and uncoupled respiratory conditions, and the maximal rate of oligomycin-sensitive ATP synthesis. In addition, to definitely establish whether patients' fibroblasts are energy deficient, intracellular ATP levels will be measured . State 4 and State 3 respiration rates will be measured in the absence and in the presence of saturating ADP, respectively, and the uncoupled respiration in the presence of the uncoupler FCCP (Carbonyl cyanide-p-trifluoromethoxyphenylhydrazone). The Complex I driven ATP synthesis rate will be measured under the state 3 respiratory conditions described above. The synthesized ATP or steady state ATP content of cells will be quantified by a luminometric method.

iv) mitochondrial dysfunction leads to mitochondrial membrane potential (MMP) changes and ROS production. Thus, MMP, a main functional parameter of mitochondria, will be estimated in cells by both fluorescence microscopy and flow cytometry to detect alterations of both the mitochondrial network and the inner mitochondrial membrane potential Δψm. Δψm will be measured by loading cells with tetramethylrhodamine methyl ester (TMRM), a lipophilic probe which enters mitochondria in a Δψm-dependent manner. Cells will be incubated with TMRM either in the absence or presence of oligomycin, a specific inhibitor of the ATP synthase complex , and under FCCP. Multiple high-power fluorescence images of patients and controls fibroblasts will be acquired by fluorescence inverted microscope using IAS2000 software (Delta Sistemi, Roma, Italy). For quantitative Δψm analysis by flow cytometry, a MUSE cell analyzer (Millipore, Billerica, MA, USA) will be used applying the Flowing software (Centre for Biotechnology, University of Turku). Any evidence of mitochondrial alterations will be further addressed by immunoblotting of OXPHOS complexes v) in parallel to in vivo assessment, the possible contribution of higher ROS level and consequent cellular oxidative stress in the pathogenesis of RFC1-ataxia will be evaluated in cultured fibroblasts, by measuring anion superoxide radical (O2 • -) mitochondrial levels by the fluorescent probe MitoSOX Red, and cellular ROS level by the CellROX Orange fluorescent probe, using a MUSE cytometer. To explore whether ROS alterations depend on changes in the antioxidant defense systems of the cells, levels and activities of the main antioxidant enzymes and total and reduced glutathione level will be assessed by immunoblot and spectrophotometric assays, respectively.

vi) the finding of significant mitochondrial alterations in RFC1 fibroblasts will prompt to investigate their proneness to mitochondrial-induced cell death. Increased ROS induces permeability transition of the cyclosporine-sensitive pore in the inner mitochondrial membrane, which in turn causes mitochondria swelling and consequent disruption of both ATP synthesis and ion homeostasis, leading to cell death. Apoptosis activation will be assessed in patient and control cells in glucose enriched-DMEM medium at different times. Proneness to cell death will be evaluated by the Muse cell analyzer using the Muse Count and viability assay Kit, Annexin V and Dead Cell Assay Kit, and Caspase-3/7 Assay Kit.

As last additional aim, in this study, iPSCs will be established. Three RFC1 and three controls PF culture lines will be induced into iPSCs , in collaboration/supervising with dr J Rosati, IRCCS Casa Sollievo della Sofferenza. These IPSc will be further differentiated into primary proprioceptive neurons, as sensory neurons result invariably affected in RFC1-ataxia patients.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of RFC1-ataxia
* age >18 years and <80 years
* ability to sign informed consent

Exclusion Criteria:

* Diagnosis of other degenerative and/or non-degenerative neurological diseases
* Not signed informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) scale | 1 year
  SARA is a clinical scale validated in degenerative ataxias, which assesses a range of different impairments related to cerebellar dysfunction. The scale is made up of 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test ; Each item scores from 0 ( no impairment) to 4 ( maximum impairment) Global SARA score ranges from 0 (no cerebellar ataxia ) to 40 (maximal severity of ataxia )
INTERNATIONAL CO-OPERATIVE ATAXIA RATING SCALE (ICARS) | 1 year
  ICARS is another, recommended outcome scale for cerebellar ataxias, including 19 items and 4 subscales evaluating postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders (14); Each subscale has an ordinal scale with 0 indicating normal and the higher score indicating greatest impairment or that the patient is unable to complete the task. Global score ranges from 0 to 100 : higher score indicates greater impairment
SENSORY ATAXIA RATING SCALE (SEARS) | 1 year
  SEARS is a 10-item functional scale developed and validated to cover the clinical spectrum of manifestations in patients with sensory neuronopathies. It has been validated for any forms of sensory ataxia, including 10-meter walking test (10mWT) to assess gait speed. Scores range from 0 (no impairment) to 41 (maximal impairment)
Berg Balance Scale (BBS) | 1 year
  BBS for balance assessment is an ordinal scale ranging from 0 to 56, consisting of 13 items with a score from 0 to 4 where 0 is the minimum performance and 4 is the maximum performance regarding the item required. This scale mainly evaluates the static balance and minimally the dynamic
Tinetti scale | 1 year
  The Tinetti Assessment Tool is a simple test that measures both gait and balance abilities based on performing specific tasks. Scoring of the Tinetti Assessment Tool is done on a 3-point ordinal scale with a range of 0 to 2, where 0 represents the most impairment, while 2 represents independence. The individual scores are then combined to form three measures: an overall gait assessment score (maximum score 12), overall balance assessment score (maximum score 16), combined gait and balance score (maximum total score is 28). Scores below 19 indicate high risk for falls
Dizziness Handicap Inventory Scale (DHI) | 1 year
  The DHI evaluates the self-perception of the incapacitating effects, on the quality of life, caused by dizziness. It comprises 25 items with a total score ranging between 0 and 100 points. DHI can be further subdivided into physical (DHI-P, 28 points), functional (DHI-F 36 points) and emotional (DHI-E 36 points) sub scores. A higher score indicates a more severe handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Silvestri, Principal Investigator — Catholic University of the Sacred Heart
Locations (2):
- Italy (2):
  - Alma Mater Studiorum University of Bologna, Bologna
  - Department of Neuroscience, Roma